CLINICAL TRIAL: NCT05718453
Title: Assessment of Trace Elements, Systemic Inflammation and Electrolytes in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Assessment of Trace Elements, Systemic Inflammation and Electrolytes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rasha Abdelfattah
Record Dates: First submitted 2023-01-04; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Copd
Keywords: COPD; Biomarkers; Trace elements; Electrolytes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Intervention Model Description: Measurement of serum level of CRP, tumor necrosis factor, zinc, copper, potassium, sodium, and magnesium in patients with stable COPD and during exacerbation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPD patients (Active Comparator): It is about 60 patients with Stable COPD
  Interventions: Combination Product: Laboratory Tests
- Acute exacerbation COPD (Active Comparator): It is about 40 patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD).
  Interventions: Combination Product: Laboratory Tests
- healthy controls (Placebo Comparator): It is about 40 healthy controls were included in the study
  Interventions: Combination Product: Laboratory Tests

INTERVENTIONS:
Combination Product: Laboratory Tests — Measurement of serum level of CRP, tumor necrosis factor, zinc, copper, potassium, sodium, and magnesium in patients with stable COPD and during exacerbation.

SUMMARY:
COPD is one of the most common causes of health problems worldwide. It is a disease that is associated with several systemic features that affect its morbidity and mortality.

DETAILED DESCRIPTION:
The most prominent features of COPD are systemic inflammation and oxidative stress. There is growing interest in establishing the significance of systemic inflammatory biomarkers in COPD patients, as they could be useful in evaluating exacerbations, monitoring disease progression, and evaluating treatment outcomes.

C-reactive protein (CRP) is a biomarker for systemic inflammation, produced mostly by hepatocytes in response to tissue injury or inflammation.

Tumor necrosis factor - alpha (TNF-α) is a key modulator of the immune system's response to infection. At the sites of inflammation, this cytokine regulates the function of poly-morphs and lymphocytes, with essentially protective benefits for the host. Increased TNF-α production may enhance an injury process locally and also elevated circulating levels may have negative systemic consequences.

Trace elements are hypothesized to play a role in the pathogenesis of many diseases, either directly or indirectly. Trace elements play an important function in the inhibition and activation of enzyme processes .

Zinc, for example, is a co-factor for various enzymes and is important for cell membrane stability, protein synthesis, proper tissue growth, and nucleic acid metabolism.

Severity of COPD exacerbation is associated with increased levels of copper (Cu) and zinc (Zn).

Patients with COPD are liable for various electrolyte derangements, especially during exacerbations. Hyponatremia is typically observed in the final stages of COPD. Hypokalemia may also occur independently or concomitantly with hyponatremia, and because magnesium plays a role in muscle tone, a drop in magnesium levels in COPD is a component that reduces respiratory muscle function and causes muscle fatigue.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients

Exclusion Criteria:

* Patients with Cardiovascular diseases,
* diabetes mellitus,
* chronic kidney disease,
* chronic liver disease,
* collagen vascular diseases,
* cancer,
* currently smoking,
* current pneumonia or inflammation, or refused to participate in the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the pain resulted in COPD | from baseline to 72 hours
  The Pain was measured by using the visual analogue score (VAS) as Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain
Number of participants with abnormal laboratory test results | from baseline to 48 hours after the taking blood samle
  he study tried to assess some Laboratory Tests in blood and comparing the level of their results in patients with stable and patients with exacerbation of theirs disease and aslo comparing their values between patients who needed and those who did not need mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad O Abdel Aziz, Professor, Study Director — Department of Internal medicine Minia university, Minia, Egypt
Locations (1):
- Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No